CLINICAL TRIAL: NCT03049891
Title: Impact of Decentralization on Retention of Pediatric Patients Initiated on ART at a Large Referral Hospital in Eastern Cape, South Africa
Brief Title: Pediatric Decentralization of ART in South Africa
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Elaine J. Abrams, MD, Research Director, ICAP at Columbia University, Columbia University
Other Study IDs: AAAO9854
Record Dates: First submitted 2017-02-06; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: HIV/AIDS
Keywords: Antiretroviral Therapy; Retention; Loss to Follow Up
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Children down-referred from DNH: This group includes children who were transferred from DNH to a study facility. The investigators will first abstract data from the electronic data system 'Tier.net' for these children, which will tell us where they were down-referred. For children who were labeled as down-referred from DNH in Tier.net, data abstraction of the child's clinical data will be conducted at the down-referral site and from the National Health Laboratory Service (NHLS) data.
  Interventions: Other: Data abstraction; Other: Tier.net
- Children LTF from DNH: This group includes children who began ART at DNH and were subsequently LTF. The investigators will first abstract data from the electronic data system 'Tier.net', which will classify them as LTF followed by examination of the the NHLS laboratory data to determine whether these children had received care at another facility since they were LTF.
  Interventions: Other: Data abstraction; Other: Tier.net
- Caregivers of LTF: This group includes the caregivers of a subset of children in the 'LTF from DNH' and 'down-referred from DNH' groups. Among those children down-referred and LTF from DNH, the investigators will use their clinical and laboratory data to determine whether they are still receiving care or not. For children identified as LTF based on their abstracted data will be traced in order to contact their caregivers. If located, caregivers will be interviewed to ascertain if and why these children are no longer in care through a 'Tracing questionnaire'.
  Interventions: Other: Tracing questionnaire
- DNH only: This group includes children who are still in care at DNH, died while in care at DNH, or were transferred to facilities from tier.net will not have any additional information collected other than what is recorded in the Tier.net database.
  Interventions: Other: Tier.net

INTERVENTIONS:
Other: Data abstraction — The investigators will abstract clinical data from down-referral sites and from NHLS to determine whether children made it to their down-referral sites or whether children are in care at a different facility.
  Other Names: NHLS (National Health Laboratory Service)
  Groups: Children LTF from DNH; Children down-referred from DNH
Other: Tracing questionnaire — The investigators will attempt to contact and visit caregivers of children who are determined to be LTF from DNH or from down-referral sites. If located and after providing consent, caregivers will be administered a tracing questionnaire, or a verbal autopsy if their child has died.
  Groups: Caregivers of LTF
Other: Tier.net — For all children who started ART at DNH between 2004 and 2013, the investigators will abstract data on these children from the electronic medical system in South Africa called Tier.net.
  Groups: Children LTF from DNH; Children down-referred from DNH; DNH only

SUMMARY:
The decentralization study will describe children taking antiretroviral therapy (ART) at a larger health facility in the Eastern Cape province of South Africa, between the years of 2004-2013. The study will be conducted at Dora Nginza Hospital (DNH). The study will measure how many children stay in care and how many die, as well as their health status. The study will also compare whether children do better if they stay in care a large hospitals or if they get health care at smaller clinics. A second part of the study will find children in the community who have stopped coming for health care and find out what happened to them and what their health status is.

DETAILED DESCRIPTION:
The investigators propose to conduct a two part study which will include a retrospective cohort study to examine care outcomes among pediatric patients 0-14 years of age initiated on antiretroviral therapy (ART) in 2004-2013 at a larger peri-urban health facility in the Eastern Cape province of South Africa. The study will be conducted at Dora Nginza Hospital (DNH). The outcomes measured in the study will include retention and mortality, as well as virologic suppression rates for children initiated on ART. In addition to reporting outcomes for all children with available data, the study will compare outcomes for children retained in care at DNH (where they initiated ART) to those children who were referred out after initiation for routine follow-up at community health clinics and primary care clinics ("down referred"). A second part of the study will trace pediatric patients in the community who have been lost to follow-up (LTF) to ascertain their outcomes after they left care at the health facility.

ELIGIBILITY:
ART Outcomes Study:

Inclusion Criteria:

* HIV positive; less than 15 years of age; started ART at DNH between 2004 and 2013.

Exclusion Criteria:

* Anyone not meeting inclusion criteria

Tracing Study:

Inclusion Criteria:

* Legal caregiver (older than 18) a child who was included in the ART Outcomes Study that was found to be LTFU from DNH or from the down-referral facility.

Exclusion Criteria:

* Guardians who cannot be confirmed as the legal caregiver of the child

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study consists of two parts. The first part is a retrospective records review of electronic and medical records of children starting ART at a large hospital facility 2004-2013 (no sampling or recruitment). We expect that 1600 children started ART during this period. The second part of the study will be a community tracing study of children who have been lost to follow-up, in which we will interview caregivers of children. We will randomly sample 75 patients who have been LTF will be generated using the data from the retrospective records review.
Sampling Method: Non-Probability Sample
Enrollment: 1583 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children initiated on ART at DNH who are still in care | Baseline (single measure)

SECONDARY OUTCOMES:
Proportion of children with hospitalization and/or death after ART initiation at DNH | Baseline (single measure)
Proportion of down-referred children retained in care at their down-referral facility. | Baseline (single measure)
Proportion of children who died or were LTF among those who remained at DNH and those down-referred | Baseline (single measure)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine J Abrams, MD, Principal Investigator — ICAP at Columbia University
Locations (15):
- South Africa (15):
  - Chatty Clinic, Port Elizabeth, Eastern Cape
  - Dora Nginza Hospital, Port Elizabeth, Eastern Cape
  - Empilweni TB Hospital, Port Elizabeth, Eastern Cape
  - Govan Mbeki Clinic, Port Elizabeth, Eastern Cape
  - Joe Slovo Clinic, Port Elizabeth, Eastern Cape
  - Kwadwesi Clinic, Port Elizabeth, Eastern Cape
  - Kwazakhele Clinic, Port Elizabeth, Eastern Cape
  - Kwazakhele Community Health Center, Port Elizabeth, Eastern Cape
  - Motherwell Community Health Center, Port Elizabeth, Eastern Cape
  - New Brighton Clinic, Port Elizabeth, Eastern Cape
  - New Brighton Community Health Center, Port Elizabeth, Eastern Cape
  - Soweto Clinic, Port Elizabeth, Eastern Cape
  - Walmer 14th Avenue Clinic, Port Elizabeth, Eastern Cape
  - West End Clinic, Port Elizabeth, Eastern Cape
  - Zwide Clinic, Port Elizabeth, Eastern Cape